CLINICAL TRIAL: NCT05457920
Title: The Efficacy and Safety of IHCs Treated With Pegylated Interferon α2b Based on Pulse Theray or Sequential Therapy
Brief Title: Study on Clinical Program Optimization of Inactive Hepatitis B Surface Antigen (HBsAg) Carriers (IHCs)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanPPHGRS
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Chronic Hepatitis B
Keywords: inactive hepatitis B virus carriers; Pegylated Interferon α2b; Continuous treatment, pulse treatment
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (continuous treatment group) (Experimental): The treatment period is 12 weeks as a treatment unit, starting from the first day of baseline, subcutaneous injection of Peg-IFNα-2b 180μg once a week, the total treatment course does not exceed 96 weeks. During treatment, when any efficacy check point reaches the disappearance of HBsAg with or without the appearance of HBsAb, at least 2 treatment units of consolidation therapy are given and then the drug is discontinued. Observed for 24 weeks after treatment.
  Interventions: Behavioral: continuous treatment
- Group B (pulse therapy group) (Experimental): The treatment period is 12 weeks as a treatment unit. From the first day of baseline, subcutaneous injection of Peg-IFNα-2b 180 μg, every injection for 8 weeks, stop for 4 weeks, periodically, the total treatment course does not exceed 96 weeks. During treatment, when any efficacy check point reaches the disappearance of HBsAg with or without the appearance of HBsAb, at least 2 treatment units of consolidation therapy are given and then the drug is discontinued. Observed for 24 weeks after treatment.
  Interventions: Behavioral: pulse therapy

INTERVENTIONS:
Behavioral: continuous treatment — The treatment period is 12 weeks as a treatment unit, starting from the first day of baseline, subcutaneous injection of Peg-IFN α-2b 180μg once a week, or every 8 weeks of injection, 4 weeks off, periodically, the total treatment course does not exceed 96 weeks.
  Arms: Group A (continuous treatment group)
Behavioral: pulse therapy — pulse therapy
  Arms: Group B (pulse therapy group)

SUMMARY:
A multicenter, randomized controlled trial design was used to select patients with chronic hepatitis B in the immune control phase (i.e. HBsAg positive, HBeAg negative, normal ALT and HBsAg≤1000IU/ml, HBV DNA≤2000IU/ml) to enter this study, and to compare the feasibility, effectiveness and safety treated with Pegylated Interferon α2b Continuous therapy or Pulse therapy in immune-controlled chronic hepatitis B patients.

DETAILED DESCRIPTION:
Patients:chronic hepatitis B in the immune control phase (i.e. HBsAg positive, HBeAg negative, normal ALT and HBsAg≤1000IU/ml, HBV DNA≤2000IU/ml). The study patients were divided into two groups.Group A (PEG IFN α- 2b continuous group): PEG IFN was injected subcutaneously once a week from the first day of baseline α- 2b 180 μg. The total course of treatment should not exceed 96 weeks.Group B (PEG IFN α- 2b pulse group): from the first day of baseline, PEG IFN was injected subcutaneously α- 2b 180 μg. Every 8 weeks of injection, stop for 4 weeks, and conduct it periodically.Two groups at baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72weeks, 84 weeks, 96 weeks and the 12th and 24th weeks after drug withdrawal, and corresponding examinations were carried out at each follow-up.Check and record adverse events and concomitant medication in detail, and evaluate the compliance of subjects; Blood samples were retained and transported to the laboratory for HBV at baseline, 24 weeks, 48weeks, 72, 96, and 12 and 24 after drug withdrawal.DNA quantification and detection of hepatitis B virus markers.The efficacy and safety were evaluated after the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years, both male and female (including 18 and 65 years old);
* HBV DNA≤2000 IU/ml and HBeAg negative;
* HBsAg positive for more than 6 months, and HBsAg≤1000 IU/ml;
* ALT≤ULN at screening (discontinue liver-protecting enzyme-lowering drugs for at least 2 weeks);
* A negative urine or serum pregnancy test (for women of childbearing age) within 24 hours before the first dose;
* B-ultrasound or fibroscan suggest no liver cirrhosis;
* Willing to accept treatment and sign informed consent.

Exclusion Criteria:

* Participants with other hepatotropic viruses or human immunodeficiency virus co-infection;
* other chronic non-viral liver diseases or decompensated liver diseases;
* tumours;
* drug abuse;
* severe psychiatric disease;
* uncontrolled thyroid disease or diabetes;
* pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Extent of HBsAg decrease at 48 weeks | 48 weeks
  Decreasing level and difference of HBsAg in different treatment groups after 48 week treatment

SECONDARY OUTCOMES:
HBsAg clearance at the end of 96 weeks of treatment | 96 weeks
  To determine the response rate will be evaluated by HBsAg loss defined as HBsAg level lower than 0.05 IU/ml after 96 week treatment
The decreasing extent of HBsAg level at 96 weeks | 96 weeks
  Decreasing level and difference of HBsAg in different treatment groups after 96 week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shang, Study Chair — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
After publication
Supporting Information: Study Protocol
Time Frame: End of study
Access Criteria: Editors and reviewers of contributing magazines